CLINICAL TRIAL: NCT05979389
Title: Pilot Trial of Bicalutamide Versus Placebo in Reproductive-Aged Women With Nonalcoholic Fatty Liver Disease (NAFLD) and Polycystic Ovary Syndrome (PCOS)
Brief Title: Bicalutamide Therapy in Young Women With NAFLD and PCOS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 23-39274; R01DK134633-01A1 (NIH)
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: NAFLD; PCOS
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — bicalutamide

STUDY DESIGN:
Intervention Model Description: The following treatment regimens will be used:
  * Experimental treatment - bicalutamide, 50 mg once daily
  * Placebo or Comparator - one capsule, once daily
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the objectives of the study, the identity of test and control treatments will not be known to investigators, research staff, or patients. The following study procedures will be in place to ensure double-blind administration of study treatments Access to the randomization code will be strictly controlled. A color and size-matched placebo capsule that looks identical to the bicalutamide capsule will be used.
  Packaging and labeling of test and control treatments will be identical to maintain the blind.
  The study blind will be broken on completion of the clinical study, after all study endpoints have been ascertained by blinded study coordinators and after the study database has been locked.
  During the study, the blind may be broken only in emergencies when knowledge of the patient's treatment group is necessary for further patient management. The University of California San Francisco investigational pharmacy would then be notified and responsible for unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bicalutamide (Experimental): 50 mg capsule administered orally once daily for 6 months
  Interventions: Drug: Bicalutamide 50 mg
- Placebo (Placebo Comparator): Matching placebo capsule administered orally once daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bicalutamide 50 mg — Bicalutamide capsules will be prepared from U.S. Pharmacopeia grade powder at a dose of 50 mg
  Other Names: Casodex
  Arms: Bicalutamide
Drug: Placebo — Matching placebo capsules of the same color, mass, and appearance to the bicalutamide capsules will be filled using microcrystalline cellulose powder.
  Arms: Placebo

SUMMARY:
Nonalcoholic steatohepatitis (NASH), or fat-related liver inflammation and scarring is projected to be the leading cause of cirrhosis in the United States (U.S.) within the next few years. Women are at disproportionate risk for NASH, with approximately 15 million U.S. women affected. There is an urgent need to understand risk factors for NASH and its progression in women, and sex hormones may provide a missing link. This study will study the contribution of androgens to liver injury and progression in PCOS and mechanistic role of dysregulated lipid metabolism and visceral adiposity in this process. Such findings will provide the rationale for future efficacy studies evaluating selective androgen receptor (AR) antagonism for NASH in PCOS, or alternatively, the need to directly target visceral adiposity or lipid-specific pathways as part of a precision medicine approach to halt fibrosis progression in the nearly 5 million young women with PCOS and NAFLD in the U.S., who remain at increased risk for early onset and progressive liver disease.

DETAILED DESCRIPTION:
This is a single center, double-blind, placebo-controlled, randomized, (1:1) parallel group pilot clinical trial of bicalutamide in women with either biopsy-proven or believed NAFLD receiving 6 months of bicalutamide or placebo. 50 women are targeted for enrollment. Each participant will be administered a single dose of bicalutamide or placebo once daily for a total of 6 months. In person evaluations will take place at Month 1, 2, 3, 4, 5, and 6. There will be a telephone follow up visit within 1 month of end of treatment. This is a pilot clinical trial that is largely feasibility focused. Study outcomes will include:

* Change in liver stiffness on Magnetic Resonance Elastography (MRE)
* Change in hepatic steatosis by Magnetic Resonance Proton Density Fat Fraction (PDFF)
* Change in visceral adipose tissue (VAT) volume by Magnetic Resonance Imaging (MRI)
* Change in NASH histology as assessed by the continuous NAFLD activity score (NAS), which measures different components of NASH on liver biopsy.
* Biochemical endpoints: serum lipids & HOMA-IR
* Feasibility outcomes including Rates (and reasons) for the following: a) % women that decline/women contacted for study inclusion (i.e. concern regarding randomization to placebo) b) % women enrolled/women screened (i.e. exclusion criteria too narrow), c) study dropout (i.e. medication side effects, too frequent study visits, and/or phlebotomy)

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-42 years with hyperandrogenic PCOS
* NASH identified on liver biopsy or probable NASH on transient elastography- controlled attenuation parameter (TE-CAP) with cutoffs defined as CAP score ≥270 decibel/m and TE score > 7.0 kPA or alanine aminotransferase ≥40 U/L).

Exclusion Criteria:

* Uncontrolled diabetes
* Alcohol consumption >2 drinks per day for at least 3 consecutive months over the previous 5 years
* Other chronic liver disease (i.e. hepatitis B virus, hepatitis C virus, autoimmune hepatitis) or cirrhosis from any cause
* Recent or planned upcoming weight reduction surgery within five years of diagnosis of biopsy-confirmed NASH
* HIV infection
* Drugs associated with fatty liver (i.e. amiodarone, methotrexate, systemic glucocorticoids, tamoxifen, anabolic steroids, valproic acid) for more than 4 weeks prior to baseline or during study
* Recent, current, or planned upcoming pregnancy or current perimenopausal status
* Renal impairment (glomerular filtration rate <45 ml/min/1.73m or potassium levels > 5.0 mmol/L)
* Androgen receptor antagonist use (i.e. spironolactone or flutamide) for more than 3 months within one year prior to baseline

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in liver stiffness on Magnetic Resonance Elastography (MRE) | Baseline and 6 months
  The investigators will assess for change in the MRE quantified liver stiffness in kilopascals (kPA)

SECONDARY OUTCOMES:
Change in hepatic steatosis by Magnetic Resonance Proton Density Fat Fraction (PDFF) | Baseline and 6 months
  The investigators will assess for percent change in fat fraction by MRI-PDFF
Change in visceral adipose tissue (VAT) volume by Magnetic Resonance Imaging (MRI) | Baseline and 6 months
  The investigators will assess for percent change in VAT as quantified by MRI
Change HOMA-IR (Homeostatic model assessment (HOMA) for insulin resistance (IR)) | Baseline and 6 months
  The investigators will assess change in continuous measures of HOMA-IR as insulin resistance is known to contribute to NASH progression
Change in the NAFLD Activity Score (NAS) on a scale from 0 (low activity) to 8 (high activity) | Baseline and 6 months
  The investigators will assess for change in this histologic scoring system of NASH as a continuous measure among women willing to undergo end of treatment biopsy (not required).

CONTACTS AND LOCATIONS:
Overall Officials: Monika A Sarkar, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maldonado SS, Grab J, Wang CW, Huddleston H, Cedars M, Sarkar M. Polycystic ovary syndrome is associated with nonalcoholic steatohepatitis in women of reproductive age. Hepatol Commun. 2022 Oct;6(10):2634-2639. doi: 10.1002/hep4.2039. Epub 2022 Jul 21. PMID 35861548
- [Background] Sarkar MA, Suzuki A, Abdelmalek MF, Yates KP, Wilson LA, Bass NM, Gill R, Cedars M, Terrault N; NASH Clinical Research Network. Testosterone is Associated With Nonalcoholic Steatohepatitis and Fibrosis in Premenopausal Women With NAFLD. Clin Gastroenterol Hepatol. 2021 Jun;19(6):1267-1274.e1. doi: 10.1016/j.cgh.2020.09.045. Epub 2020 Oct 1. PMID 33010412
- [Background] Sanchez-Garrido MA, Tena-Sempere M. Metabolic dysfunction in polycystic ovary syndrome: Pathogenic role of androgen excess and potential therapeutic strategies. Mol Metab. 2020 May;35:100937. doi: 10.1016/j.molmet.2020.01.001. Epub 2020 Feb 5. PMID 32244180
- [Background] O'Reilly MW, Kempegowda P, Walsh M, Taylor AE, Manolopoulos KN, Allwood JW, Semple RK, Hebenstreit D, Dunn WB, Tomlinson JW, Arlt W. AKR1C3-Mediated Adipose Androgen Generation Drives Lipotoxicity in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2017 Sep 1;102(9):3327-3339. doi: 10.1210/jc.2017-00947. PMID 28645211
- [Background] Dieudonne MN, Pecquery R, Boumediene A, Leneveu MC, Giudicelli Y. Androgen receptors in human preadipocytes and adipocytes: regional specificities and regulation by sex steroids. Am J Physiol. 1998 Jun;274(6):C1645-52. doi: 10.1152/ajpcell.1998.274.6.C1645. PMID 9611130
- [Background] Gambineri A, Patton L, Vaccina A, Cacciari M, Morselli-Labate AM, Cavazza C, Pagotto U, Pasquali R. Treatment with flutamide, metformin, and their combination added to a hypocaloric diet in overweight-obese women with polycystic ovary syndrome: a randomized, 12-month, placebo-controlled study. J Clin Endocrinol Metab. 2006 Oct;91(10):3970-80. doi: 10.1210/jc.2005-2250. Epub 2006 Jul 25. PMID 16868063
- [Background] Cusi K. Role of obesity and lipotoxicity in the development of nonalcoholic steatohepatitis: pathophysiology and clinical implications. Gastroenterology. 2012 Apr;142(4):711-725.e6. doi: 10.1053/j.gastro.2012.02.003. Epub 2012 Feb 8. PMID 22326434
- [Background] Macut D, Tziomalos K, Bozic-Antic I, Bjekic-Macut J, Katsikis I, Papadakis E, Andric Z, Panidis D. Non-alcoholic fatty liver disease is associated with insulin resistance and lipid accumulation product in women with polycystic ovary syndrome. Hum Reprod. 2016 Jun;31(6):1347-53. doi: 10.1093/humrep/dew076. Epub 2016 Apr 12. PMID 27076501
- [Background] Kumarendran B, O'Reilly MW, Manolopoulos KN, Toulis KA, Gokhale KM, Sitch AJ, Wijeyaratne CN, Coomarasamy A, Arlt W, Nirantharakumar K. Polycystic ovary syndrome, androgen excess, and the risk of nonalcoholic fatty liver disease in women: A longitudinal study based on a United Kingdom primary care database. PLoS Med. 2018 Mar 28;15(3):e1002542. doi: 10.1371/journal.pmed.1002542. eCollection 2018 Mar. PMID 29590099
- [Background] Ismail FF, Meah N, Trindade de Carvalho L, Bhoyrul B, Wall D, Sinclair R. Safety of oral bicalutamide in female pattern hair loss: A retrospective review of 316 patients. J Am Acad Dermatol. 2020 Nov;83(5):1478-1479. doi: 10.1016/j.jaad.2020.03.034. Epub 2020 Mar 22. No abstract available. PMID 32213304
- [Background] Fernandez-Nieto D, Saceda-Corralo D, Rodrigues-Barata R, Hermosa-Gelbard A, Moreno-Arrones O, Jimenez-Cauhe J, Ortega-Quijano D, Vano-Galvan S. Oral bicalutamide for female pattern hair loss: A pilot study. Dermatol Ther. 2019 Nov;32(6):e13096. doi: 10.1111/dth.13096. Epub 2019 Oct 10. No abstract available. PMID 31579984